CLINICAL TRIAL: NCT06720792
Title: An Escape Game to Promote Students' Mental Health Outcomes in the Aftermaths of Covid-19 Pandemic: Protocol for a Randomized Controlled Trial Evaluating a Cocreated Intervention
Brief Title: Cocreation and Evaluation of an Escape Game on Students' Mental Health
Acronym: EscapeCovid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bordeaux (Other)
Collaborators: David Labrosse (Unknown); Clara Vié (Unknown)
Responsible Party: Principal Investigator, Montagni Ilaria, Lecturer-researcher, University of Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANR-21-CE36-0011; ANR-21-CE36- 0011-02 (Other: Agence Nationale de Recherche)
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Mental Health
Keywords: cocreation; evaluation; randomised controlled trial; students; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game play (Active Comparator): Participants receive an email with the link to book a slot to play the Escape Game. The date when students can play the Escape Game is defined when 4 students are available at the same slot. Students receive a further email with all the instructions to play the game.
  Interventions: Other: EscapeCovid
- email on mental health-related information (Placebo Comparator): Students receive an email detailing mental health services and describing the most common mental health problems. Participants are randomized so that the two groups are similar in terms of sex, age and field of study (stratified balanced randomization).
  Interventions: Other: EscapeCovid

INTERVENTIONS:
Other: EscapeCovid — Online Escape Game with 4 players and a game guide. The players, in a group, must solve enigmas to win.

SUMMARY:
The Covid-19 pandemic and the protracted lockdowns have heavily impacted university students' mental health. Digital Escape Games represent a good means to reach students and propose them solutions for their psychological well-being.

The objective of the study is to evaluate a cocreated digital Escape Game on students' mental health in the Covid-19 era. The evaluation of the effectiveness of this stand-alone intervention concerns mental health outcomes (mental health literacy, appraisal and change of beliefs about mental health, recognition and management of emotions, and positive coping strategies) and the appreciation and relevance of the game.

A randomized controlled trial with pre- and post-test data collection (online questionnaires with validated scales) will be conducted among 500 students in Bordeaux, France, to evaluate a game cocreated with students, researchers, health professionals and web-developers. A sub-sample of students will be randomly selected for responding to a semi-structured interview following a mixed methods design. Recruitment will be done through mail invitation from student associations and presentations in university classes. Half of the sample (250 students) will play the Escape Game, while the other half will receive an email with mental health-related information. The whole study is carried out online.

As of December 2nd 2024, 191 students have answered the baseline questionnaire (90 intervention vs. 101 control). Twenty-three students have played the Escape Game and 53 are in the control arm. The current sample size is too small for reaching significance level. Among participants, 20 were interviewed (10 intervention vs. 10 control) reaching the saturation of the sample. According to preliminary results, the game has proved a positive impact on all defined outcomes, while the email has been effective in increasing knowledge on resources available and on coping strategies and meditation techniques. We expect the trial to be completed by the end of June 2025.

Preliminary results from the qualitative sub-study are promising: in the aftermaths of the Covid-19 crisis, this intervention is intended to promote players' mental health through gamification, knowledge transfer and a learning-by-doing approach.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate through a randomized controlled trial and semi-structured interviews (mixed methods design) an intervention on mental health promotion and on psychological disease prevention in the form of a digital Escape Game addressed to University students in the era of Covid-19.

The specific objectives of the study are:

1. assessing among students the effectiveness of the digital Escape Game in (a) increasing players' mental health literacy, (b) helping appraise and change students' beliefs about mental health, (c) supporting recognition and management of their emotions, and (d) teaching them useful positive coping strategies;
2. assessing the impact of the digital Escape Game on participants' levels of anxiety, stress and depression; and
3. questioning the appreciation and relevance of the digital Escape Game among students.

Consequential research hypotheses of the study are:

1. compared to the control group receiving another intervention, after playing the digital Escape Game, students have remarkably improved the following mental health indicators: mental health literacy, identification and positive change of beliefs about mental health, recognition and management of emotions, and adoption of positive coping strategies;
2. the intervention group also presents reduced levels of anxiety, depression and stress after having played the game one week, one month and three months after the intervention (comparison with the control group and within the group); and
3. digital Escape Games are considered as appealing and relevant by students when treating mental health.

The Escape Game will be evaluated through a rigorous Randomized Controlled Trial (RCT) design using pre- and post-intervention data coming from a repeated online self-administered questionnaire. The investigators will compare the answers between exposed and non-exposed students (inter-group) and measure the change in their answers at three timepoints (intra-group). The investigators will recruit at least 500 students at the University of Bordeaux, France (this number has been confirmed with a statistical power calculation targeting participants in each arm to achieve 80% to 90% power to detect a small effect - f = 0.09 to f = 0.10 - for differential change in the 2 arms, with α = .05.) representative of the student population in Bordeaux for sex, year and field of study, according to the statistics of the University of Bordeaux. Students will be invited through posts on the social media of the study partners and mailing lists from the University of Bordeaux. Inclusion criteria are: being a student in Bordeaux, being aged ≥18 years and having given the electronic consent to participate to the study (check the "I agree" box to be enrolled in the study, after having read its conditions). After having signed the consent form, students can access the baseline questionnaire. Based on the completion of the questionnaires, the recruitment will end once the sample is composed of at least 500 students (this will be checked by a continuous monitoring through descriptive analysis). At the end of the baseline questionnaire, participants will be allocated to either the intervention or the control group through a random assignment. Thus, 250 students will play online the Escape Game, while 250 students will receive an email with tips and resources for managing their stress during the Covid-19 pandemic. Participants will be randomized so that the two groups are similar in terms of sex, age and field of study (stratified balanced randomization).

Briefly, the 250 students of the intervention arm will: (1) complete the baseline questionnaire, (2) play the Escape Room within the week after the baseline questionnaire, and (3) complete the same questionnaire of the baseline at three timepoints, i.e. one week, one month and three months after having played the game (follow-up). The 250 students of the control arm will: (1) complete the baseline questionnaire, (2) receive the same day an email with tips and resources to manage their stress during the Covid-19 pandemic, and (3) complete the same questionnaire of the baseline at three time points, i.e. one week, one month and three months after having received the email.

In the questionnaire sent after one week after having played the game, the intervention group will also have to respond to some items on the appreciation of the game (satisfaction survey). All participants will be rewarded with gift cards to maximize recruitment and follow-up (the gift card will be offered after the third follow-up at month 3).

Following a mixed methods design, 20 students will be randomly selected among the 250 having received the intervention to respond to a semi-structured interview. Data from these interviews is about commenting on the perceived improvement of the mental health indicators of the quantitative phase and about appreciation and relevance of the intervention. The sample will be composed in order to have different profiles, so that 20 is an approximative number of participants that could be higher or lower depending on the sample saturation. The interviews will be conducted based on an ad hoc grid, transcribed and analyzed through triangulation.

The questionnaires will include validated scales measuring mental health literacy (the Mental Health Literacy Scale - MHLS), health-related beliefs (the Health Belief Model - HBM), emotions (the Differential Emotions Scale - DES), coping strategies (the Ways of Coping strategy Questionnaire - WCQ), anxiety (Generalized Anxiety Disorder-7 (GAD-7), depression (Patient Health Questionnaire-9, (PHQ-9)) and stress (Perceived Stress Scale-4 (PSS-4)).

The items on appreciation/relevance of the intervention will be created ad hoc, but will also be inspired by existing instruments evaluating digital health interventions.

The final questionnaire will be developed by several researchers through different stages of drafts and reviews, following a structured survey construction method in 5 steps.

The response modalities will be varied: multiple choice, binary responses, Likert scales and visual analogue scales. Mental health indicators and appreciation/relevance results are the main outcomes of the study.

Analysis and interpretation of the data will follow the mixed methods approach: first, statistical analyses on quantitative data (descriptive statistics, modeling, exploratory data analysis); second, the discourse analysis of qualitative data (thematic analysis based on a pre-defined interview guide); and third, the coupled analysis of both types of data according to the explanatory design procedure. According to this procedure, qualitative data are used to explain the quantitative results.

ELIGIBILITY:
Inclusion Criteria:

* university students
* understanding and speaking French
* being aged more than 18 years old

Exclusion Criteria:

* not enrolled in a French university
* minor
* not understanding and speaking French
* not having given one's electronic consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Mental Health Literacy Scale | Up to 3 months (baseline + one week + one month and three months after having played the Escape Game or having received the email.the email
  Validated scale on knowledge, information and beliefs about mental health. Score range from 35 to 160. There are no categories, it is a continuous score.
The Health Belief Model Scale | Up to 3 months (baseline + one week + one month and three months after having played the Escape Game or having received the email. Score ranges from 1 to 5, continuous variable.
  Validated scale on how we perceive and represent health in general and mental health in particular
The Differential Emotions Scale | Up to 3 months (baseline + one week + one month and three months after having played the Escape Game or having received the email.the email
  Validated scale for assessment of an individual's emotions. Mean, standard deviation, variance.
The Ways of Coping strategy Questionnaire | Up to 3 months (baseline + one week + one month and three months after having played the Escape Game or having received the email.the email
  Validated questionnaire describing one's resilience and knowledge of strategies to promote (mental) health and prevent (mental) diseases
Acceptability and relevance of the game | One week after having played the Escape Game or having received the email.
  Ad hoc items to describe the appreciation of the game. Sum of the answers, continuous variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux Population Health U1219, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided
De-identified participant data will be available from the principal investigator upon request, exclusively after the conclusion of the trial.

REFERENCES:
- [Background] Vie C, Govindin-Ramassamy K, Thellier D, Labrosse D, Montagni I. Effectiveness of digital games promoting young people's mental health: A review of reviews. Digit Health. 2024 Feb 5;10:20552076231220814. doi: 10.1177/20552076231220814. eCollection 2024 Jan-Dec. PMID 38323239
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Plutchik R. The measurement of emotions. Acta Neuropsychiatr. 1997 Jun;9(2):58-60. doi: 10.1017/S0924270800036802. PMID 26972127
- [Background] Montagni I, Gonzalez Caballero JL. Validation of the Mental Health Literacy Scale in French University Students. Behav Sci (Basel). 2022 Jul 28;12(8):259. doi: 10.3390/bs12080259. PMID 36004830
- [Background] Janz NK, Becker MH. The Health Belief Model: a decade later. Health Educ Q. 1984 Spring;11(1):1-47. doi: 10.1177/109019818401100101. PMID 6392204
- [Background] Aschentrup L, Steimer PA, Dadaczynski K, Mc Call T, Fischer F, Wrona KJ. Effectiveness of gamified digital interventions in mental health prevention and health promotion among adults: a scoping review. BMC Public Health. 2024 Jan 2;24(1):69. doi: 10.1186/s12889-023-17517-3. PMID 38167010
- [Background] Arrue M, Suarez N, Ugartemendia-Yerobi M, Babarro I. Let's play and learn: Educational escape room to improve mental health knowledge in undergraduate nursing students. Nurse Educ Today. 2025 Jan;144:106453. doi: 10.1016/j.nedt.2024.106453. Epub 2024 Oct 11. PMID 39418755
- [Result] Labrosse D, Vie C, Hajjam H, Tisseron C, Thellier D, Montagni I. An Escape Game on University Students' Mental Health During the COVID-19 Pandemic: Cocreation Study. JMIR Serious Games. 2024 Mar 18;12:e48545. doi: 10.2196/48545. PMID 38498033
- [Derived] Labrosse D, Vie C, Harb M, Montagni I. Escape Game to Promote Students' Mental Health Outcomes in the Aftermaths of COVID-19 Pandemic: Protocol for a Mixed Methods Study Evaluating a Cocreated Intervention. JMIR Res Protoc. 2025 Apr 2;14:e64068. doi: 10.2196/64068. PMID 40173436